CLINICAL TRIAL: NCT03100825
Title: A Multicenter, Open-label, Single Arm, 52-week Treatment Study to Assess the Safety of QVM149 in Japanese Patients With Asthma
Brief Title: A Long-term Safety Study of QVM149 in Japanese Patients With Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CQVM149B1304
Record Dates: First submitted 2017-03-29; First posted 2017-04-04 (Actual); Results first posted 2020-04-07 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-03

CONDITIONS: Asthma
Keywords: QVM149; Asthma; Japanese; Allergic asthma; Allergy triggered asthma; Reactive asthma; Asthma attack; Difficulty breathing
MeSH Terms: conditions — Asthma; Dyspnea | interventions — Parturition; Powders; Hardness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QVM149 (Experimental): All eligible patients take QVM149 150/50/160 μg once daily over 52 weeks.
  Interventions: Drug: QVM149

INTERVENTIONS:
Drug: QVM149 — QVM149 (indacaterol acetate/glycopyrronium bromide/mometasone furoate)
  Other Names: QVM149 150/50/160 μg once daily, delivered as powder in hard capsules via Concept1 inhaler

SUMMARY:
The purpose of this study is to provide long term safety data of QVM149 in Japanese patients with asthma for the registration of QVM149 in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained before any assessment is performed.
* Male and female adult patient ≥ 18 years old.
* Patients with a diagnosis of persistent asthma (GINA 2016) for a period of at least 1 year prior to Visit 1.
* Patients who have used medium or high dose of ICS/LABA combinations for asthma for at least 3 months and at stable dose and regimen for at least 4 weeks prior to Visit 1.
* An ACQ-7 score ≥ 1.5 at Visits 2.
* Pre-bronchodilator FEV1 of ≥ 40% and ≤ 85% of the predicted normal value for the patient after withholding bronchodilators at Visit 2.

  o Repeating is allowed once only. Repeating of percentage predicted FEV1 should be done in an ad-hoc visit to be scheduled on a date that would provide sufficient time to receive confirmation from the spirometry data central reviewer of the validity of the assessment before Visit 99.
* Patients must demonstrate reversibility defined as an increase in FEV1 of ≥ 12% and 200 mL within 15 to 30 minutes after administration of 400 µg of salbutamol at Visit 2. Spacer devices are permitted during reversibility testing only. The Investigator or delegate may decide whether or not to use a spacer for the reversibility testing.

  * If reversibility is not proven at Visit 2, patients may be permitted to enter the study with historical evidence of reversibility that was performed within 5 years prior to Visit 1.
  * Alternatively, patients may be permitted to enter the study with a historical positive bronchoprovocation test (defined as a provoked fall in FEV1 of 20% by bronchoconstriction agent e.g., methacholine, histamine) or equivalent test (e.g., astography) that was performed within 5 years prior to Visit 1.
  * If reversibility is not proven at Visit 2 and historical data is not available, reversibility should be repeated once in an ad-hoc visit scheduled as close as possible from the first attempt (but not on the same day).

Exclusion Criteria:

* Patients who have had an asthma attack/exacerbation requiring systemic steroids or hospitalization or emergency room visit within 6-weeks of Visit 1.
* Patients who have ever required intubation for a severe asthma attack/exacerbation.
* Patients who have a clinical condition which is likely to be worsened by ICS administration (e.g. glaucoma, cataract and fragility fractures) who are according to investigator's medical judgment at risk participating in the study.
* Patients with narrow-angle glaucoma, symptomatic benign prostatic hyperplasia (BPH) or bladder-neck obstruction or severe renal impairment or urinary retention. BPH patients who are stable on treatment can be considered.
* Patients who have had a respiratory tract infection or asthma worsening as determined by investigator within 4 weeks prior to Visit 1 or between Visit 1 and Visit 99. Patients may be re-screened 4 weeks after recovery from their respiratory tract infection or asthma worsening.
* Patients with a history of chronic lung diseases other than asthma, including (but not limited to) COPD, sarcoidosis, interstitial lung disease, cystic fibrosis, clinically significant bronchiectasis and active tuberculosis.
* Patients with severe narcolepsy and/or insomnia
* Pregnant or nursing (lactating) women
* Women of child-bearing potential unless they are using highly effective methods of contraception during dosing and for 30 days after stopping of investigational medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2017-04-28 (Actual); Primary Completion 2018-09-18 (Actual); Study Completion 2019-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (21):
- Japan (21):
  - Novartis Investigative Site, Koga, Fukuoka
  - Novartis Investigative Site, Yanagawa, Fukuoka
  - Novartis Investigative Site, Maebashi, Gunma
  - Novartis Investigative Site, Hiroshima, Hiroshima
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Tomakomai, Hokkaido
  - Novartis Investigative Site, Takamatsu, Kagawa-ken
  - Novartis Investigative Site, Fujisawa, Kanagawa
  - Novartis Investigative Site, Sagamihara, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Yokkaichi, Mie-ken
  - Novartis Investigative Site, Nagaoka, Niigata
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Sakai, Osaka
  - Novartis Investigative Site, Ageo, Saitama
  - Novartis Investigative Site, Chuo Ku, Tokyo
  - Novartis Investigative Site, Chuo-ku, Tokyo
  - Novartis Investigative Site, Ōta-ku, Tokyo
  - Novartis Investigative Site, Setagaya-ku, Tokyo
  - Novartis Investigative Site, Shinagawa-ku, Tokyo
  - Novartis Investigative Site, Toshima Ku, Tokyo

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 161 participants were screened, of which 94 participants entered the treatment phase. A total of 86 participants completed the study.
Groups:
- QVM149: Participants received QVM149 (indacaterol acetate/glycopyrronium bromide/mometasone furoate) 150/50/160 micrograms (mcg) once daily as powder in hard capsules via Concept1 inhaler in the evening throughout treatment epoch of 52 weeks.
Period: Overall Study
Arm/Group | QVM149
Started | 94
Completed | 86
Not Completed | 8
Not completed — Participant/Guardian Decision | 7
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Groups:
- QVM149: Participants received QVM149 (indacaterol acetate/glycopyrronium bromide/mometasone furoate) 150/50/160 mcg once daily as powder in hard capsules via Concept1 inhaler in the evening throughout treatment epoch of 52 weeks.
Arm/Group | QVM149
Number analyzed (Participants) | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (12.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 94
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  East Asian | 94
Height [Mean (Standard Deviation); unit: Centimeters (cm)] | 164.17 (8.495)
Weight [Mean (Standard Deviation); unit: Kilogram (kg)] | 68.31 (14.044)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kilograms per meter square (kg/m^2)] | 25.29 (4.554)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs)
Description: An adverse event (AE) was any untoward medical occurrence (example; any unfavorable and unintended sign including abnormal laboratory findings, symptom or disease) in a participant or clinical investigation participant after providing written informed consent for participation in the study until the end of study visit. TEAEs were defined as adverse events started on or after the time of the first inhalation of study drug but no later than 7 days after the last administration (30 days in the case of SAEs). SAE was defined as any adverse event (appearance of [or worsening of any pre-existing]) undesirable sign, symptom or medical conditions which is fatal or life-threatening or results in persistent or significant disability/incapacity or constitutes a congenital anomaly/birth defect or requires inpatient hospitalization or prolongation of existing hospitalization or is medically significant.
Time Frame: Up to 52 Weeks
Population: Safety set included all participants who received at least one dose of study medication during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | QVM149
Number analyzed (Participants) | 94
Participants
  TEAEs | 64
  SAEs | 6

2. Secondary Outcome: Change From Baseline (Pre-dose) Forced Expiratory Volume in One Second (FEV1) at Week 26 and 52
Description: FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation, measured through spirometry testing. Change from baseline in FEV1 at week 26 and 52 was reported.
Time Frame: Baseline (Pre-dose), Week 26, Week 52
Population: Full Analysis Set (FAS) included all participants who entered in the treatment epoch of this study and received at least one dose of study medication during the study. Here, 'n' (number analyzed) signified number of participants evaluable for specified time points.
Measure: Mean (Standard Deviation); unit: Liters (L)
Arm/Group | QVM149
Number analyzed (Participants) | 94
Liters (L)
  Week 26: number analyzed (Participants) | 83
  Week 26 | 0.3789 (0.34896)
  Week 52: number analyzed (Participants) | 80
  Week 52 | 0.3598 (0.38878)

3. Secondary Outcome: Change From Baseline (Pre-dose) Forced Vital Capacity (FVC) at Week 26 and 52
Description: Forced Vital Capacity is the amount of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. FVC was assessed by spirometry. Change from baseline in FVC at week 26 and 52 was reported.
Time Frame: Baseline (Pre-dose), Week 26, Week 52
Population: FAS included all participants who entered in the treatment epoch of this study and received at least one dose of study medication during the study. Here, 'n' (number analyzed) signified number of participants evaluable for specified time points.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | QVM149
Number analyzed (Participants) | 94
L
  Week 26: number analyzed (Participants) | 83
  Week 26 | 0.2938 (0.35997)
  Week 52: number analyzed (Participants) | 80
  Week 52 | 0.2860 (0.42054)

4. Secondary Outcome: Change From Baseline in Morning and Evening Peak Expiratory Flow (PEF) Over 52 Weeks
Description: PEF is the peak expiratory flow, the maximum speed of expiration. Electronic peak flow meter (ePEF) was given to each participant at visit 1 for the measurement of morning and evening PEF. Change from baseline in morning and evening PEF over 52 weeks was measured.
Time Frame: Baseline up to week 52
Population: FAS included all participants who entered in the treatment epoch of this study and received at least one dose of study medication during the study. Here, 'n' (number anlayzed) signified number of participants evaluable for the specified time points.
Measure: Mean (Standard Deviation); unit: liters per minute (L/min)
Arm/Group | QVM149
Number analyzed (Participants) | 94
liters per minute (L/min)
  Morning | 42.26 (61.913)
  Evening | 35.48 (60.710)

5. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire-7 (ACQ-7) Total Score at Week 26 and 52
Description: ACQ-7 is a 7-item, disease-specific instrument developed and validated to assess asthma control in participants. All 7 items were scored on a 7-point Likert scale, with 0 indicating total control of asthma and 6 indicating poor control of asthma. The questions were equally weighted and the total score is the mean of the 7 items. A decrease of ACQ-7 score of at least 0.5 from baseline was considered to be clinically meaningful improvement.
Time Frame: Baseline, Week 26, Week 52
Population: FAS included all participants who entered in the treatment epoch of this study and received at least one dose of study medication during the study. Here, 'n' (number analyzed) signified number of participants evaluable for the specified time points.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | QVM149
Number analyzed (Participants) | 94
Score on a scale
  Week 26: number analyzed (Participants) | 89
  Week 26 | -0.881 (0.5629)
  Week 52: number analyzed (Participants) | 84
  Week 52 | -0.935 (0.6155)

6. Secondary Outcome: Proportion of Participants Who Achieved Clinically Meaningful Improvement Threshold in ACQ-7 Score (Decrease of Greater Than or Equal to 0.5 Units in ACQ-7) at Week 26 and 52
Description: ACQ-7 is a 7-item, disease-specific instrument developed and validated to assess asthma control in participants. All 7 items were scored on a 7-point likert scale, with 0 indicating total control of asthma and 6 indicating poor control of asthma. Questions were equally weighted and total score is mean of 7 items. A decrease from baseline of at least 0.5 units in ACQ-7 score was considered to be clinically meaningful improvement. The proportion of participants achieving the clinically meaningful improvement threshold in ACQ-7 score were reported at Week 26 and Week 52.
Time Frame: Week 26, Week 52
Population: Analysis population included FAS with ACQ-7 data at the respective visit. Here 'n' (number analyzed) signified number of participants evaluable for specified time points.
Measure: Number; unit: Percentage of participants
Arm/Group | QVM149
Number analyzed (Participants) | 89
Percentage of participants
  Week 26 | 67.4
  Week 52: number analyzed (Participants) | 84
  Week 52 | 73.8

7. Secondary Outcome: Change From Baseline in Daily Number of Puffs of Rescue Medication Over 52 Weeks
Description: Daily use of rescue medication (number of puffs taken in the previous 12 hours) were recorded each morning and evening throughout the 52 week treatment by the participant using their electronic diary.
Time Frame: Baseline up to week 52
Population: FAS included all participants who entered in the treatment epoch of this study and received at least one dose of study medication during the study. Here 'N' (overall number of participants analyzed) signified number of participants evaluable for the outcome measure.
Measure: Mean (Standard Deviation); unit: Number of puffs
Arm/Group | QVM149
Number analyzed (Participants) | 93
Number of puffs | -0.29 (0.895)

ADVERSE EVENTS:
Time Frame: From start of study treatment up to 52 Weeks
Description: An Adverse Event (AE) any sign or symptom that occurs during the study treatment
Groups:
- QVM149: Participants received QVM149 (indacaterol acetate/glycopyrronium bromide/mometasone furoate) 150/50/160 μg once daily in the evening throughout treatment epoch of 52 weeks.
Arm/Group | QVM149
All-Cause Mortality (participants affected / at risk) | 0/94
Serious Adverse Events (participants affected / at risk) | 6/94
Other Adverse Events (participants affected / at risk) | 57/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QVM149 (N=94)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Cataract (Eye disorders) | 1
Anal fistula (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Oesophageal rupture (Gastrointestinal disorders) | 1
Appendicitis (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Uterine leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QVM149 (N=94)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2
Pyrexia (General disorders) | 3
Acute sinusitis (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 6
Cystitis (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 2
Influenza (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 17
Pharyngitis (Infections and infestations) | 5
Rhinitis (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 2
Contusion (Injury, poisoning and procedural complications) | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Trigger finger (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 29
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 10
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3
Eczema (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2017-04-06): https://cdn.clinicaltrials.gov/large-docs/25/NCT03100825/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-06): https://cdn.clinicaltrials.gov/large-docs/25/NCT03100825/SAP_001.pdf